CLINICAL TRIAL: NCT04076449
Title: Quantitative Susceptibility Mapping Biomarker, Brain Structure and Connectome Associated With Cerebral Cavernous Malformation Related Epilepsy and Outcome After Surgery
Brief Title: Quantitative Susceptibility Biomarker and Brain Structural Property for Cerebral Cavernous Malformation Related Epilepsy
Acronym: CRESS
Status: Recruiting | Type: Observational
Sponsor: yuanli Zhao (Other)
Collaborators: Peking University International Hospital (Other)
Responsible Party: Sponsor-Investigator, yuanli Zhao, Professor, Department of Neurosurgery, Beijing Tiantan Hospital
Organization: Beijing Tiantan Hospital (Other)
Other Study IDs: KYSQ 2018-020-01; H0906 81801140 (Other Grant/Funding Number: National Nature Science Foundation)
Record Dates: First submitted 2019-08-29; First posted 2019-09-03 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-09

CONDITIONS: Cavernous Malformation, Cerebral; Cavernous Angioma; Cavernous Hemangioma; Cavernous Hemangioma of Brain; Seizures; Seizures, Epileptic; Epilepsy
Keywords: Cerebral Cavernous Malformation; Epilepsy; Quantitative Susceptibility Mapping (QSM); Brain Connectome; Cerebral Structure
MeSH Terms: conditions — Hemangioma, Cavernous, Central Nervous System; Hemangioma, Cavernous; Seizures; Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Surgical resected lesion and 20 ml blood sample before surgery
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cerebral Cavernous Malformation with Epilepsy: Patients with cerebral cavernous malformation and associated with epilepsy will undergo MR imaging and be followed-up annually as our protocol defined.
- Cerebral Cavernous Malformation without Epilepsy: Patients with cerebral cavernous malformation but without epilepsy will undergo MR imaging and be followed-up annually as our protocol defined.

SUMMARY:
Cerebral cavernous malformation (CCM)-related epilepsy (CRE) impairs the quality of life in patients with CCM. Patients could not always achieve seizure freedom after surgical resection of the lesion, suggesting an inadequate treatment and evaluation of the epileptogenic zone or network. Iron deposition in cerebral cavernous malformations has been postulated to play an important role in triggering CRE. Quantitative susceptibility mapping (QSM), as an optimal in vivo imaging technique to quantify iron deposition, is employed to analyze the iron quantity in CCM patients with epilepsy and further combined with brain structural and connectome analysis, to describe the difference between CCMs with and without epilepsy. In vivo biomarkers predicting CRE risk in CCM natural history and CRE control outcome after CCM surgical resection will be further identified to improve management strategy.

DETAILED DESCRIPTION:
The CRESS study is a prospective observational study of imaging biomarker for cerebral cavernous malformation (CCM) related epilepsy (CRE) risk in natural history or after surgical resection. This project, funded by the National Nature Science Foundation of China, will be performed in two sites: Bejing Tiantan Hospital, Capital Medical University and Peking University International Hospital, which cover the south and north part of Beijing. Bejing Tiantan Hospital is also the China National Clinical Research Center for Neurological Diseases and the largest neurological center with high volume of patients all over the nation.

Study overview: Each participants will be followed for 5 year since enrollment. Epilepsy will be tracked with serial video EEG recordings and clinical investigations performed annually. Besides medical history of the patients, data from seizure diary and MR imaging studies (including quantitative susceptibility mapping, diffusion tensor imaging and three dimension-T1 weighted imaging), will be collected. Blood samples and tissue samples of surgical resected lesion for biomarkers studies will also be collected in all participants of the project. The data obtained in participants of CCM with or without epilepsy will be compared.

Sample size: Investigators plan to enroll 200 CCM patients in 24 months and follow up for 5 years. Based upon the preliminary results and extensive literature review, investigators predict that about 50% of participants will undergo surgical treatment, while 25% of participants remain suffering from seizure after treatment.

Study endpoints: The primary clinical endpoint of this study is a collection of a set of clinical, molecular, and MRI data in all participants.

ELIGIBILITY:
Inclusion Criteria:

* (1) 18 to 70 years of age
* (2) Diagnosed with a single cerebral cavernous malformation
* (3) No prior treatment of the symptomatic lesion

Exclusion Criteria:

* (1) Associated with brain lesions and/or tumors other than CCM
* (2) History of previous intracranial surgery
* (3) Prior brain irradiation
* (4) Contraindication or unwilling or unable to undergo research MRI studies
* (5) Pregnant or breastfeeding women
* (6) Persons unable or unlikely to return for follow-up visits
* (7) Dementia or other progressive neurological disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Outpatient and inpatient referred to Beijing Tiantan Hospital and Peking University International Hospital who diagnosed with cerebral cavernous malformation.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-09-03 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Perilesional mean QSM in CCM with conservative treatment | End of study (5-year) MRI scan
  Each patient contributes five outcome measurements (at annual image of 5-year follow-up). Perilesional QSM measurements will be performed at baseline and at annual epoch of image. Perilesional mean QSM (in parts per million, ppm) in each study group will be evaluated using univariate comparison and a repeated measures analysis implemented as an unadjusted linear mixed model.
Perilesional mean QSM after surgical resection of CCM lesion | End of study (3-year) MRI scan after surgery
  Each patient contributes three outcome measurements (at year 1 and 2 and 3 after surgery). Perilesional QSM measurements will be performed at annual imaging follow-up after surgery. Mean QSM (in parts per million, ppm) in patients with or without postoperative seizure will be evaluated using univariate comparison and a repeated measures analysis implemented as an unadjusted linear mixed model.
Ratio of seizure freedom during follow-up | End of follow-up period (5-year)
  Seizure freedom, defined as Engel Classification of Post-treatment Outcome Class I, will be assessed annually during follow-up period. For patients with medical treatment or conservative observation, the follow-up period begins since enrollment. For patients with surgical resection, the follow-up period begins after surgery.

SECONDARY OUTCOMES:
Grey matter volume in CCM with epilepsy | End of study (5-year) MRI scan
  The presurgical grey matter volume will be calculated from three dimension T1 weighted imaging. Data of CCM with or without epilepsy will be compared and to detect the correlation between grey matter volume and seizure severity (Liverpool Seizure Severity Scale) and frequency.
Whole-brain connectome in CCM with epilepsy | End of study (5-year) MRI scan
  Whole-brain connectome will be reconstructed from whole-brain diffusion tensor imaging before surgical treatment. Data of CCM with or without epilepsy will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Li Ma, MD, PhD, Principal Investigator — Beijing Tiantan Hospital
Locations (2):
- China (2):
  - Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking University International Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol to be published in peer-reviewed journal
Supporting Information: Study Protocol
Time Frame: Since the publication of study protocol
Access Criteria: Available from the principle investigator upon reasonable request

REFERENCES:
- [Derived] Liu Y, Wen Z, Yuan J, Ma L, Wu C, Wu J, Liu Q, Zhang S, Wang S. Venous Architecture Predicts Hemorrhage Risk in Sporadic CCM With DVA. Stroke. 2025 Dec;56(12):3361-3370. doi: 10.1161/STROKEAHA.125.052339. Epub 2025 Sep 3. PMID 40899314
- [Derived] Ma L, Zhang S, Li Z, Wu CX, Wang Z, Zhan L, Hao Q, Wang H, Ye X, Chen X, Liu YO, Wang S, Zhao YL. Morbidity After Symptomatic Hemorrhage of Cerebral Cavernous Malformation: A Nomogram Approach to Risk Assessment. Stroke. 2020 Oct;51(10):2997-3006. doi: 10.1161/STROKEAHA.120.029942. Epub 2020 Sep 21. PMID 32951540